CLINICAL TRIAL: NCT05270772
Title: A Single-arm, Open-label Phase I Study of CAR-T-19 (Anti CD19 scFv Chimeric Antigen Receptor T) Cells for Patients With CD19-positive Recurrent or Refractory B-cell Acute Lymphoblastic Leukemia Under The Age of 25
Brief Title: CAR-T-19 Cells for Patients With CD19+ Relapse/Refractory B-ALL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Daihong Liu, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT19-ALL-02
Record Dates: First submitted 2022-02-26; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-01

CONDITIONS: CD19+ Relapse/Refractory B-ALL
Keywords: B-ALL; CAR-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T-19 Cells (Experimental): The patients with CD19+ relapse or refractory B-ALL will receive a single infusion of autologous CAR-T-19 cells, with the escalated dose ranging from 0.5×10^6/kg to 5.0×10^6/kg CAR+ cells.
  Interventions: Biological: CAR-T-19 Cells

INTERVENTIONS:
Biological: CAR-T-19 Cells — T cells were isolated from the PBMC of patients, transduced with lentivirus, expanded in vitro, and infused into patients. The escalated doses include 0.5×10^6/kg,1.5×10^6/kg, 5.0×10^6/kg CAR+ cells.

SUMMARY:
This is a single-arm, open-label phase I study to determine the safety, tolerability, and recommended dose (RD) of CAR-T-19 cells for patients with CD19+ relapse/refractory B-ALL under the age of 25.

DETAILED DESCRIPTION:
B-cell acute lymphoblastic leukemia (B-ALL) accounting for 85% of all ALL cases, is a common hematological malignancy in children and adults. CD19 is a widely expressed antigen in both normal B cells and B cells-derived leukemia and lymphomas. This is a single-arm, open-label phase I study of CAR-T-19 (anti CD19 scFv chimeric antigen receptor T) cells for patients with CD19-positive relapse/refractory B-ALL under the age of 25.

Primary endpoint is to determine the safety, tolerability, and recommended dose (RD) of CAR-T-19. Secondary endpoints measure ORR, OS and others.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapse/refractory B-ALL.
* Tumor cells from bone marrow or peripheral blood are measured CD19+ with 3 months before enrollment.
* Karnofsky Score ≥ 70 or Lansky Score ≥ 50.
* Patients who have a life expectancy of at least 12 weeks.
* Understand and voluntarily sign informed consent and are willing to comply with laboratory tests and other research procedures.

Exclusion Criteria:

* Patients with extramedullary relapse (EMR).
* Patients with genetic diseases, Burkitt lymphoma and leukemia or other malignancies.
* Patients positive for any of the following: HbsAg, HBV-DNA, HCV-Ab, HCV-RNA, HIV-Ab, TP-Ab, EBV-DNA or CMV-DNA.
* Patients with other uncontrolled infection.
* Patients who received anti-CD19 / anti-CD3 therapy, or any other anti-CD19 therapy.
* Patients with active Grade II-IV GVHD within 3 months prior to screening.
* Tumor cells are detected in cerebrospinal fluid.
* Patients who received HSCT within 3 months prior to screening.
* Anticipated other clinical trials within 4 weeks before this trial
* Pregnant or lactating women.
* Any condition that would, in the investigator's judgment, make it unsuitable for the donors to be enrolled.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2024-09-16 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | up to 2 years
  DLT within 28 days (±3 days) after CAR-T-19 infusion.
Maximum tolerated dose (MTD) | up to 2 years
  The maximum dose of DLT occurred in ≤1/6 of the subjects within 28 days (±3 days) after CAR-T-19 infusion.
Adverse events | up to 2 years
  Percentage of subjects with adverse events.

SECONDARY OUTCOMES:
Overall recovery rate (ORR) | up to 2 years
  Percentage of subjects who achieved complete response (CR) and incomplete hematologic recovery (CRi) for the first time at Day 28 and Day 90 after CAR-T-19 infusion.
MRD-Negative Rate | up to 2 years
  Percentage of subjects with MRD-negative CR and incomplete blood and MRD-negative CRi for the first time at Day 28 and Day 90 after CAR-T-19 infusion.
Duration of Response (DOR) | up to 2 years
  The time from achieving CR and CRi for the first time to recurrence or death from any cause
Progression-free Survival (PFS) | up to 2 years
  The time from CAR-T-19 infusion to recurrence, progression or death from any cause, whichever occurs first.
Overall survival (OS) | up to 2 years
  The time from CAR-T-19 infusion to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China